CLINICAL TRIAL: NCT01367496
Title: An Open-Label, Phase I Study of the Pharmacokinetics and Bioavailability of Single, Ascending Subcutaneous Doses of Methylnaltrexone Versus Intravenous Dose in Normal, Healthy Male Volunteers
Brief Title: Pharmacokinetics and Bioavailability of Single Subcutaneous Doses of Methylnaltrexone Versus Intravenous Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D., Progenics Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 103
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: SC Methylnaltrexone (MNTX)
- Arm 2 (Experimental)
  Interventions: Drug: SC Methylnaltrexone (MNTX)
- Arm 3 (Experimental)
  Interventions: Drug: SC Methylnaltrexone (MNTX)
- Arm 4 (Experimental)
  Interventions: Drug: IV Methylnaltrexone (MNTX)

INTERVENTIONS:
Drug: SC Methylnaltrexone (MNTX) — Dose 1
  Arms: Arm 1
Drug: SC Methylnaltrexone (MNTX) — Dose 2
  Arms: Arm 2
Drug: SC Methylnaltrexone (MNTX) — Dose 3
  Arms: Arm 3
Drug: IV Methylnaltrexone (MNTX)
  Arms: Arm 4

SUMMARY:
This is an open-label, Phase I study. Study treatments will entail a four-way crossover among three single, ascending, subcutaneous doses and one intravenous dose of MNTX in six healthy normal male volunteers. Blood samples will be obtained to determine plasma pharmacokinetics, dose proportionality for subcutaneous doses, and absolute bioavailability versus an intravenous dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subject weight between 60 and 80 kg
2. Subject a non-smoker
3. Subject in good physical health, based on history, physical exam, appropriate laboratory and diagnostics tests at screening with no evidence of clinically significant chronic medical condition.

Exclusion Criteria:

1. Subject with known hypersensitivity to methylnaltrexone, naltrexon or other opioids
2. Subject consuming any prescription medication within the past two weeks, over-the-counter (OTC) products within seven days, any experimental medication within 30 days prior to study screening, or of any drug with a half-life longer then three days within 10 half-lives (>30 days) of screening
3. Subject consuming barbiturates or other inducers or inhibitors of CYP450 within 3 months of screening
4. Subject with history or evidence of cardiovascular, gastrointestinal, hepatic, neurological, pulmonary, and renal or other significant chronic illness.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2002-06; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration of MNTX | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.

SECONDARY OUTCOMES:
Time to Maximum Plasma Concentration (Tmax) of MNTX | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.
Clearance of MNTX | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.
Half-live of MNTX | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.
Volume of Distribution of MNTX | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.
Area Under the Plasma Concentration versus Time Curve (AUC) of MNTX | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.
Urinary Clearance of MNTX | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.
Percentage of MNTX Excreted in Urine | 32 days
  The objective of this study is to determine the plasma pharmacokinetic of single, ascending, subcutaneous doses and a single intravenous dose of methylnaltrexone (MNTX) in normal healthy male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States